CLINICAL TRIAL: NCT02961725
Title: Umbilical Cord Mesenchymal Stem Cells for Treatment of Bronchopleural Fistula
Brief Title: Stem Cells for Treatment of Bronchopleural Fistula
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Fujian Medical University (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-BF
Record Dates: First submitted 2016-11-03; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Bronchopleural Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UCMSC treatment (Experimental): UCMSC: umbilical cord mesenchymal stem cells
  Interventions: Biological: UCMSC

INTERVENTIONS:
Biological: UCMSC — UCMSC: umbilical cord mesenchymal stem cells 3-5*10^7/5 ml

SUMMARY:
Bronchopleural fistula (BF), an abnormal passage or communication between a bronchus and another part of the body, may develop when there are penetrating wounds of the thorax and after lung surgery. Without effective therapy, treatment of BF is a challenge, with a high rate of mortality and teratogenicity.

The investigators will conduct endoscopic injection of umbilical cord mesenchymal stem cells to fistula, observe the recovery of bronchopleural fistula and systemic reactions, to investigate the application of umbilical cord mesenchymal stem cells in the treatment of bronchopleural fistula.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with bronchopleural fistula by imaging or bronchoscopic examination
* typical symptom of bronchopleural fistula, such as fever, cough, purulent sputum, weight loss…
* patients present compromised conditions, who can only accept a conservative treatment.

Exclusion Criteria:

* absolute contraindication of bronchoscopic examination and treatment
* with previous treatment of cell therapy, including stem cells.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
closure of the fistula | 24 weeks
  median time for fistula closure

SECONDARY OUTCOMES:
complication | 1 year
  fever, coughing up blood, infection...

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Zeng, Dr., Principal Investigator — The Second Affiliated Hospital of Fujian Medical University
Locations (1):
- The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided